CLINICAL TRIAL: NCT05501925
Title: GlideSheath Slender® Versus Conventional 6 French Arterial Sheath: Impact on the Incidence of Distal Radial Artery Occlusion in Cardiovascular Intervention Via Distal Radial Artery (SMART)
Brief Title: GlideSheath Slender® Versus Conventional 6 French Arterial Sheath: Impact on the Distal Radial Artery Occlusion (SMART)
Acronym: SMART
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wujin People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: WJH20220731
Record Dates: First submitted 2022-08-06; First posted 2022-08-16 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Coronary Artery Disease; Cardiovascular Diseases
Keywords: distal radial artery; distal radial artery occlusion; cardiovascular intervention
MeSH Terms: conditions — Coronary Artery Disease; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: GlideSheath Slender® group Conventional Sheath group (TERUMO, Introducer II )
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GlideSheath Slender® (Experimental): Placement of 6 French GlideSheath Slender® for cardiovascular intervention via distal radial artery
  Interventions: Device: GlideSheath Slender® and conventional arterial sheath
- Conventional Sheath (Active Comparator): Placement of 6 French conventional Sheath (TERUMO, Introducer II ) for cardiovascular intervention via distal radial artery
  Interventions: Device: Conventional arterial sheath

INTERVENTIONS:
Device: GlideSheath Slender® and conventional arterial sheath — Using the GlideSheath Slender® with the outside diameter 2.46mm
  Arms: GlideSheath Slender®
Device: Conventional arterial sheath — Placement of 6 French conventional Sheath (TERUMO, Introducer II )
  Arms: Conventional Sheath

SUMMARY:
Compared with conventional artery sheath (TERUMO, Introducer II ), GlideSheath Slender® has more smaller outer-side diameter. The investigators suspected that use of the GlideSheath Slender® can reduce the incidence of distal radial artery occlusion in cardiovascular intervention via dTRA approach.

DETAILED DESCRIPTION:
Distal transradial artery (dTRA) approach has emerged as a new approach in cardiovascular intervention in recent years. Compared to the conventional radial artery (CRA) approach, the dTRA approach dramatically reduced the risk of radial artery occlusion (RAO). In recent years, the incidence of distal radial artery occlusion (dRAO) after dTRA intervention has been reported in the literature, ranged from 0.12% to 5.2%. Outside diameter of artery sheath may affect the incidence of dRAO. Retrospective study reported that an artery/ sheath ratio > 1.0 was least damaging to the vessel during coronary intervention via dTRA. Compared with conventional artery sheath (TERUMO, Introducer II ), 6 French GlideSheath Slender® has more smaller outer-side diameter (2.46mm vs. 2.62mm). The investigators suspected that use of the GlideSheath Slender can reduce the incidence of dRAO in cardiovascular intervention via dTRA approach.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Palpable distal radial and conventional radial artery

Exclusion Criteria:

* Age ≥ 90years
* Height≥ 185cm
* ST-segment elevation myocardial infarction or Cardiogenic shock
* Contraindications to puncture at the puncture site
* Diameter of DRA less than 1.5mm or RAO

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Rate of distal radial artery occlusion | 24 hours after the coronary angiography or intervention
  The rate of distal radial artery occlusion is evaluated by ultrasound

SECONDARY OUTCOMES:
Rate of radial artery occlusion | 24 hours after the coronary angiography or intervention
  The rate of radial artery occlusion is evaluated by ultrasound
Pain during the placement of the sheath | 24 hours after the coronary angiography or intervention
  Visual analog scale is used to evaluate the pain during the placement of the sheath, which ranges from 0-10, and 0 meas no pain
Radial artery dissection | 24 hours after the coronary angiography or intervention
  The incidence of dissection of the radial artery is evaluated by ultrasound
Time of hemostasis | 24 hours after the coronary angiography or intervention
  The time from the compress to hemostasis
Haematoma | 24 hours after the coronary angiography or intervention
  The incidence of haematoma is evaluated by Early Discharge After Transradial Stenting of Coronary Arteries Study criteria

CONTACTS AND LOCATIONS:
Overall Officials: Gaojun Cai, Study Chair — Wujin hospital affiliated with Jiangsu University
Locations (1):
- Changzhou Wujin People's Hospital, Changzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kiemeneij F. Left distal transradial access in the anatomical snuffbox for coronary angiography (ldTRA) and interventions (ldTRI). EuroIntervention. 2017 Sep 20;13(7):851-857. doi: 10.4244/EIJ-D-17-00079. PMID 28506941
- [Background] Achim A, Kakonyi K, Jambrik Z, Nagy F, Toth J, Sasi V, Hausinger P, Nemes A, Varga A, Bertrand OF, Ruzsa Z. Distal Radial Artery Access for Coronary and Peripheral Procedures: A Multicenter Experience. J Clin Med. 2021 Dec 20;10(24):5974. doi: 10.3390/jcm10245974. PMID 34945269
- [Background] Tsigkas G, Papageorgiou A, Moulias A, Kalogeropoulos AP, Papageorgopoulou C, Apostolos A, Papanikolaou A, Vasilagkos G, Davlouros P. Distal or Traditional Transradial Access Site for Coronary Procedures: A Single-Center, Randomized Study. JACC Cardiovasc Interv. 2022 Jan 10;15(1):22-32. doi: 10.1016/j.jcin.2021.09.037. Epub 2021 Dec 15. PMID 34922888
- [Background] Liang C, Han Q, Jia Y, Fan C, Qin G. Distal Transradial Access in Anatomical Snuffbox for Coronary Angiography and Intervention: An Updated Meta-Analysis. J Interv Cardiol. 2021 Jul 22;2021:7099044. doi: 10.1155/2021/7099044. eCollection 2021. PMID 34381321
- [Background] Cai G, Huang H, Li F, Shi G, Yu X, Yu L. Distal transradial access: a review of the feasibility and safety in cardiovascular angiography and intervention. BMC Cardiovasc Disord. 2020 Aug 5;20(1):356. doi: 10.1186/s12872-020-01625-8. PMID 32758150
- [Background] Naito T, Sawaoka T, Sasaki K, Iida K, Sakuraba S, Yokohama K, Sato H, Soma M, Okamura E, Harada T, Yoshimachi F. Evaluation of the diameter of the distal radial artery at the anatomical snuff box using ultrasound in Japanese patients. Cardiovasc Interv Ther. 2019 Oct;34(4):312-316. doi: 10.1007/s12928-018-00567-5. Epub 2019 Jan 7. PMID 30617776
- [Derived] Li F, Zhou T, Fan X, Chen T, Shi G, Li L, Cai G. Safety and Efficacy of Distal Transradial Access in Patients With Small Diameter Distal Radial Artery: A Post Hoc Analysis of 2 Randomized Trials. Can J Cardiol. 2025 Dec 30:S0828-282X(25)01616-2. doi: 10.1016/j.cjca.2025.12.048. Online ahead of print. PMID 41478549
- [Derived] Lu W, Chen T, Wang H, Yang A, Li L, Shi G, Xue S, Li F, Xiao J, Gu J, Zhang L, Liang X, Li W, Cai G. Comparison of the Effect of a 6-French Glidesheath Slender and a Conventional Sheath on Distal Radial Artery Occlusion: A Randomized Controlled Trial. Can J Cardiol. 2024 Nov;40(11):2292-2300. doi: 10.1016/j.cjca.2024.07.011. Epub 2024 Jul 19. PMID 39032557